CLINICAL TRIAL: NCT04452955
Title: An Open Label, Multicenter, Safety and Efficacy Phase 2 Study of PRL3-Zumab in Solid Tumors
Brief Title: A Study to Assess Safety and Efficacy of PRL3-Zumab in Patients With Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-IMMUSG Pte Ltd (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 226688
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: PRL-3; Tumor; Efficacy; Safety; Pharmacokinetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRL3-zumab (Experimental): All patients will receive PRL3-zumab until clinical progression per RECIST v1.1 and iRECIST criteria, or unacceptable toxicity, or withdraws consent.
  Interventions: Biological: PRL3-zumab

INTERVENTIONS:
Biological: PRL3-zumab — Starting dose of 6 mg/kg will be administered as IV infusion over 60 minutes every 2 weeks (±2 days)

SUMMARY:
This is a multi-center, Phase 2, open-label, single dose level study of PRL3-zumab monotherapy in patients with unresectable or metastatic solid tumor.

DETAILED DESCRIPTION:
The study consists of a Screening Period (Day - 14 to Day -1), a Treatment Period during which visits will occur every 2 weeks, an End of Treatment visit within 14 days of the decision to discontinue treatment for any reason, and a Safety Follow-up visit at 14 ± 4 days after the last dose of study treatment. PRL3-zumab will be administered by intravenous (IV) infusion till patient meets any of the discontinuation criteria (progressive disease, clinically or per RECIST v1.1 and iRECIST, intolerable toxicity or withdrawal of consent). One cycle of treatment will be 4 weeks (2 infusions, 12 days ±2 days apart).

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic solid tumors willing to provide signed informed consent.
* Histopathological diagnosis and metastatic status cancer at study entry.
* Must have received at least 1 prior line of systemic therapy for metastatic disease but no more than 3 prior lines of treatment for metastatic disease.
* Life expectancy of more than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score or less than 2.
* Adequate organ and hematological function.
* Measurable disease by RECIST v1.1 and iRECIST.

Exclusion Criteria:

* Patient has known untreated or symptomatic central nervous system metastasis.
* Patient is receiving systemic glucocorticoids or other immunosuppressive treatments for autoimmune disease or any other medical condition.
* Patient has experienced a severe hypersensitivity reaction to another monoclonal antibody.
* Patient has received treatment with any systemic anti-cancer therapies within 3 weeks prior to starting study treatment.
* Patient has undergone radiotherapy ≤ 4 weeks prior to starting study treatment.
* Patient has received > 3 lines of prior systemic chemotherapy for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From first dose of study drug until disease progression or end of treatment, whichever comes first
  PFS is defined as the time from the initiation of study treatment to the date of disease progression as per RECIST v1.1 and iRECIST criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: From first dose of study drug until disease progression or end of treatment, whichever comes first.
  Description: ORR is defined as the percentage of patients with complete response (CR) or partial response (PR) as per RECIST v1.1 and iRECIST criteria from time of initiation of study treatment.
Clinical benefit rate (CBR) | Time Frame: From first dose of study drug until disease progression or end of treatment, whichever comes first
  Description: CBR is defined as the percentage of patients with CR, PR, or stable disease (SD) as per RECIST v1.1 and iRECIST criteria based on Investigator's assessment.
Overall survival (OS) | Time Frame: From first dose of study drug until disease progression or end of treatment, whichever comes first
  Description: OS is defined as the time from the initiation of study treatment to death from any cause.
Duration of response | Time Frame: From first dose of study drug until disease progression or end of treatment, whichever comes first
  Description: Duration of response is defined as the time from the initial documented response (CR or PR) to the first documented sign of disease progression as per RECIST v1.1 and iRECIST criteria or death.
Terminal elimination half life (t½) | Pre-dose and during first dose of C1, pre dose C1D15, C2D1, C2D15, C3D1, and pre dose and during the second dose of C3, pre-dose C4D1, C5D1, C6D1 and at end of treatment (up to approximately 6 months). Duration of 1 cycle is 4 weeks. C = Cycle, D = Day.
  To assess PK after single and multiple dose administration of PRL3-zumab.
Maximum plasma PRL3-zumab concentration (Cmax) | Pre-dose and during first dose of C1, pre dose C1D15, C2D1, C2D15, C3D1, and pre dose and during the second dose of C3, pre-dose C4D1, C5D1, C6D1 and at end of treatment (up to approximately 6 months). Duration of 1 cycle is 4 weeks. C = Cycle, D = Day.
  To assess pharmacokinetics (PK) after single and multiple dose administration of PRL3-zumab.
Time of Cmax (tmax) | Pre-dose and during first dose of C1, pre dose C1D15, C2D1, C2D15, C3D1, and pre dose and during the second dose of C3, pre-dose C4D1, C5D1, C6D1 and at end of treatment (up to approximately 6 months). Duration of 1 cycle is 4 weeks. C = Cycle, D = Day.
  To assess PK after single and multiple dose administration of PRL3-zumab.
Area under the concentration time curve from pre-dose (AUCinf) | Pre-dose and during first dose of C1, pre dose C1D15, C2D1, C2D15, C3D1, and pre dose and during the second dose of C3, pre-dose C4D1, C5D1, C6D1 and at end of treatment (up to approximately 6 months). Duration of 1 cycle is 4 weeks. C = Cycle, D = Day.
  To assess PK after single and multiple dose administration of PRL3-zumab.
Number of patients with adverse events and serious adverse events | From first dose of study drug until disease progression or end of treatment, whichever comes first
  To assess safety of PRL3-zumab in patients with unresectable or metastatic solid tumors.
European Quality-5D (EQ-5D) | From first dose of study drug until disease progression or end of treatment, whichever comes first
  The system comprises 5 questions, 1 for each of 5 domains: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each is rated according to 3 response levels ("no problems," "some problems," or "extreme problems").
European Organization for Research and Treatment of Cancer-quality of life quantionnaire-C30 (EORTC-QLQ-C30) | From first dose of study drug until disease progression or end of treatment, whichever comes first
  Health-related quality of life is measured by EORTC-QLQ-C30, a 30 item questionnaire. This scale consists of functioning scales and symptom scales. For functioning scales higher scores suggest better functioning; for symptom scales higher scores suggest higher symptom burden.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - HonorHealth Research, Scottsdale, Arizona
  - St. Jude Medical Center, Fullerton, California
  - The Angeles Clinic, Los Angeles, California
  - Norton Healthcare, Louisville, Kentucky
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada

REFERENCES:
- [Derived] Park DJ, Thura M, Chiu VK, Vicuna B, Ang KH, Sanchez B, Chia PL, Kuan KY, Li J, Zhang K, Zheng WH, Hsien Ng MC, Zeng Q. The PRL3-zumab paradigm: A multicenter, single-dose-level phase 2 basket clinical trial design of an unconventional cancer immunotherapy. Cell Rep Med. 2025 May 20;6(5):102120. doi: 10.1016/j.xcrm.2025.102120. Epub 2025 May 8. PMID 40345181